CLINICAL TRIAL: NCT02409667
Title: Long Term Clear Skin Maintenance Treatment Optimization in Patients With Moderate to Severe Chronic Plaque Psoriasis: A Randomized, Multicenter, Open-label With Blinded-assessment, Comparative, 52 Week Study to Evaluate the Efficacy, Safety and Tolerability of Secukinumab 300 mg s.c.
Brief Title: Plaque Psoriasis Efficacy and Safety With Secukinumab
Acronym: OPTIMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A3302
Record Dates: First submitted 2015-03-31; First posted 2015-04-07 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-02

CONDITIONS: Plaque Psoriasis
Keywords: plaque, psoriasis
MeSH Terms: conditions — Plaque, Amyloid; Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Secukinumab 300mg in PASI 90 responders (every 4 weeks) (Active Comparator): Participants with moderate to severe plaque psoriasis who had reached PASI 90 response after 24 weeks of treatment with secukinumab 300 mg subcutanous (s.c.) every 4 weeks were treated with Secukinumab 300 mg subcutanous (s.c.) from week 24 until Week 52 every 4 weeks.
  Interventions: Biological: Secukinumab
- Secukinumab 300mg in PASI 90 responders (longer intervals) (Experimental): Participants with moderate to severe plaque psoriasis who had reached PASI 90 response after 24 weeks of treatment with secukinumab 300 mg subcutanous (s.c.) every 4 weeks were treated with Secukinumab 300 mg subcutanous (s.c.) from week 24 until Week 52 every 6 weeks.
  Interventions: Biological: Secukinumab
- Secukinumab 300mg in PASI 75-90 responders (every 4 weeks) (Experimental): Participants with moderate to severe plaque psoriasis who had reached PASI 75 to <90 response after 24 weeks of treatment with secukinumab 300 mg subcutanous (s.c.) every 4 weeks will be treated with Secukinumab 300 mg subcutanous (s.c.) from week 24 until Week 52 every 4 weeks.
  Interventions: Biological: Secukinumab
- Secukinumab 300mg in PASI 75-90 responders (shorter intervals) (Active Comparator): Participants with moderate to severe plaque psoriasis who had reached PASI 75 to <90 response after 24 weeks of treatment with secukinumab 300 mg subcutanous (s.c.) every 4 weeks were treated with Secukinumab 300 mg subcutanous (s.c.) from week 24 until Week 52 every 2 weeks.
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: Secukinumab — Secukinumab for s.c. injection was supplied in single boxes each containing 2 pre-filled syringes (PFS) of 150 mg secukinumab in a 1 mL liquid formulation. Each 300 mg dose was administered as 2 PFS injections of 150 mg secukinumab.

SUMMARY:
To demonstrate in the patient pool of PASI 90 responders at Week 24 that secukinumab 300 mg s.c. when administered at a longer dosing interval is non-inferior to secukinumab 300 mg s.c. every 4 weeks treatment with respect to maintaining a PASI 90 response rate at Week 52.

ELIGIBILITY:
Main Inclusion Criteria:

1. Chronic plaque-type psoriasis diagnosed for at least 6 months prior to Screening and candidate for systemic therapy.
2. Moderate to severe psoriasis at Baseline as evidenced by:

   * PASI ≥ 10 and
   * IGA mod 2011 score of 3 or higher (based on a scale of 0 to 4) and
   * BSA affected by plaque-type psoriasis of ≥ 10%.

Main Exclusion Criteria:

1. History of exposure to any biologic drug taken for the treatment of chronic plaque psoriasis or any other indication including but not limited to anti-tumor necrosis factor (TNF) alpha, anti interleukin (IL)12/23, or any anti-IL 17A or IL 17A receptor (IL 17AR) antibody.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
3. Forms of psoriasis other than chronic plaque-type (eg, pustular, erythrodermic and guttate psoriasis).
4. Drug-induced psoriasis (ie, new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium).
5. Ongoing use of prohibited psoriasis treatments (eg, topical or systemic corticosteroids, ultraviolet (UV) therapy).
6. Ongoing use of other non-psoriasis prohibited treatments. Washout periods detailed in the protocol have to be adhered to. All other prior non-psoriasis concomitant treatments must be at a stable dose as detailed in the protocol before initiation of study drug.
7. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL).
8. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study drug and for 16 weeks after stopping study drug.
9. Active ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of secukinumab therapy.
10. Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions) which, in the opinion of the Investigator, significantly immunocompromises the patient and/or places the patient at unacceptable risk for receiving an immunomodulatory therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16487 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (170):
- Austria (3):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Loverval
- Bulgaria (6):
  - Novartis Investigative Site, Sofia, BGR
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Varna
- Croatia (3):
  - Novartis Investigative Site, Ivanić-Grad
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Zagreb
- Czechia (5):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Ostrava Poruba, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Arhus C
  - Novartis Investigative Site, Hellerup
- Finland (2):
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (12):
  - Novartis Investigative Site, Le Mans, Cedex 09
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Trévenans
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (21):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pommelsbrunn
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
- Greece (4):
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hungary (6):
  - Novartis Investigative Site, Kecskemét, Bács-Kiskun county
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Israel (5):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Roma, RM
- Latvia (4):
  - Novartis Investigative Site, Daugavpils, LVA
  - Novartis Investigative Site, Riga, LVA
  - Novartis Investigative Site, Ventspils, LVA
  - Novartis Investigative Site, Riga
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda, LTU
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Vilnius
- Netherlands (8):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Almere Stad
  - Novartis Investigative Site, Bergen op Zoom
  - Novartis Investigative Site, Geldrop
  - Novartis Investigative Site, Leiderdorp
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, Voorburg
- Poland (8):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Ossy
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (5):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Nova de Gaia
- Russia (5):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov on Don Region
  - Novartis Investigative Site, Saint Petersburg
- Slovakia (5):
  - Novartis Investigative Site, Bojnice
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Svidník
- Spain (36):
  - Novartis Investigative Site, Villajoyosa, Alicante
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, Mallorca, Mallorca
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Castellon, Valencia
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Huesca
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Pontevedra
  - Novartis Investigative Site, Zaragoza
- Sweden (4):
  - Novartis Investigative Site, Falun
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Switzerland (4):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- United Kingdom (8):
  - Novartis Investigative Site, Canterbury, Kent
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Cliftonville, Northampton
  - Novartis Investigative Site, Cannock, Staffordshire
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Harrogate

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening period was up to 4 weeks and rescreening was allowed for an unlimited number of times. At the Screening Visit, every patient was registered in an Interactive Response Technology and the Investigator ensured that the patient fulfilled all the inclusion/exclusion criteria
Groups:
- Treatment Period 1: All Participants: Participants received secukinumab 300 mg subcutaneous (s.c.) every 4 weeks for 24 weeks.
- Treatment Period 2: Group 1: Participants with moderate to severe plaque psoriasis who had reached PASI 90 response after 24 weeks of treatment with secukinumab 300 mg s.c. every 4 weeks were treated with Secukinumab 300 mg s.c. from week 24 until Week 52 every 4 weeks.
- Treatment Period 2: Group 2: Participants with moderate to severe plaque psoriasis who had reached PASI 90 response after 24 weeks of treatment with secukinumab 300 mg s.c. every 4 weeks were treated with Secukinumab 300 mg s.c. from week 24 until Week 52 every 6 weeks.
- Treatment Period 2: Group 3: Participants with moderate to severe plaque psoriasis who had reached PASI 75 to <90 response after 24 weeks of treatment with secukinumab 300 mg s.c. every 4 weeks will be treated with Secukinumab 300 mg s.c. from week 24 until Week 52 every 4 weeks.
- Treatment Period 2: Group 4: Participants with moderate to severe plaque psoriasis, who had reached PASI 75 to <90 response after 24 weeks of treatment with secukinumab 300 mg s.c. every 4 weeks, were treated with Secukinumab 300 mg s.c. from week 24 until Week 52 every 2 weeks.
Period: Treatment Period 1, Baseline to Week 24
Arm/Group | Treatment Period 1: All Participants | Treatment Period 2: Group 1 | Treatment Period 2: Group 2 | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Started | 1647 | 0 | 0 | 0 | 0
Completed | 1526 | 0 | 0 | 0 | 0
Not Completed | 121 | 0 | 0 | 0 | 0
Not completed — Withdrawal of informed consent | 6 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 20 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 5 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 48 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 25 | 0 | 0 | 0 | 0
Period: Treatment Period 2, Week 24 to Week 52)
Arm/Group | Treatment Period 1: All Participants | Treatment Period 2: Group 1 | Treatment Period 2: Group 2 | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Started | 0 | 644 | 662 | 114 | 93
Completed | 0 | 621 | 641 | 106 | 90
Not Completed | 0 | 23 | 21 | 8 | 3
Not completed — Lost to Follow-up | 0 | 7 | 4 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 7 | 4 | 1 | 2
Not completed — Withdrawal of informed consent | 0 | 5 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 5 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set for Treatment Period 1 includes all subjects who took at least one dose of study treatment during this treatment period.
Arm/Group | Treatment Period 1: All Participants
Number analyzed (Participants) | 1647
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 476
  Male | 1171
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1597
  More than one race | 0
  Unknown or Not Reported | 30

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of PASI 90 Response at Week 52 in Participants With a PASI 90 Response at Week 24
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: Week 52
Population: Full analysis set for Treatment Period 2 of PASI 90 responders (FAS-P90R): The FAS-P90R included all participants who were rated as PASI 90 responders at the Week 24 visit, randomized to treatment groups 1 or 2 and received at least one dose of study drug at or after visit Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 644 | 662
Participants | 552 | 496
Statistical Analysis 1: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Test type: Non-Inferiority — The statistical null-hypothesis to be rejected in the primary analysis was that the odds ratio of maintaining a PASI 90 response for patients with secukinumab 4-weekly dosing versus patients on secukinumab 6-weekly dosing exceeds the non-inferiority margin of 1+δ; p = 0.1499, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.44 to 2.55]

2. Secondary Outcome: Key Secondary: PASI 90 Response Rate at Week 52 in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: as for outcome 1
Time Frame: Week 52
Population: FAS for Treatment Period 2 of PASI 75 responders who did not achieve a PASI 90 response (FAS-P75R): All participants who were rated as PASI 75 responders but did not achieve a PASI 90 response at the Week 24 visit, were randomized to treatment groups 3 or 4 and who received at least one dose of study drug at or after visit Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 114 | 92
Participants | 53 | 52
Statistical Analysis 1: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Test type: Superiority; p = 0.1013, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.35 to 1.10]

3. Secondary Outcome: PASI 50, PASI 75, PASI 100 and IGA Mod 2011 0 or 1 Responders at Week 52 in Participants With a PASI 90 Response at Week 24
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50, 75, 90 and 100 were defined as participants achieving ≥ 50%, 75%, 90% or 100% improvement from baseline. The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: week 52
Population: Only participants from the FAS-P90R with evaluable data were analyzed. The FAS-P90R included all participants who were rated as PASI 90 responders at the Week 24 visit, randomized to treatment groups 1 or 2 and received at least one dose of study drug at or after visit Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 644 | 662
Participants
  PASI 50: number analyzed (Participants) | 610 | 629
  PASI 50 | 608 | 624
  PASI 75: number analyzed (Participants) | 610 | 629
  PASI 75 | 597 | 588
  PASI 90: number analyzed (Participants) | 610 | 629
  PASI 90 | 553 | 496
  PASI 100: number analyzed (Participants) | 610 | 629
  PASI 100 | 378 | 305
  IGA mod 2011: number analyzed (Participants) | 609 | 628
  IGA mod 2011 | 564 | 529

4. Secondary Outcome: PASI 50, PASI 75, PASI 100 and IGA Mod 2011 0 or 1 Responders at Week 52 in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: as for outcome 3
Time Frame: Week 52
Population: Only participants from the FAS-P75R with evaluable data were analyzed. FAS-P75R: All participants who were rated as PASI 75 responders but did not achieve a PASI 90 response at the Week 24 visit, were randomized to treatment groups 3 or 4 and who received at least one dose of study drug at or after visit Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 104 | 90
Participants
  PASI 50 | 98 | 88
  PASI 75 | 74 | 80
  PASI 90 | 53 | 52
  PASI 100 | 12 | 13
  IGA mod 2011 0 or 1 | 64 | 72

5. Secondary Outcome: Change From Baseline in PASI in Participants With a PASI 90 Response at Week 24
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). A negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 28, 32, 36, 40, 44, 48 and 52
Population: Only participants from the FAS-P90R, who had evaluable data at both baseline and the post-baseline time point, were analyzed. The FAS-P90R included all participants who were rated as PASI 90 responders at the Week 24 visit, randomized to treatment groups 1 or 2 and received at least one dose of study drug at or after visit Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 644 | 662
score on a scale
  Week 28: number analyzed (Participants) | 642 | 656
  Week 28 | -20.7 (8.471) | -19.9 (8.511)
  Week 32: number analyzed (Participants) | 638 | 655
  Week 32 | -20.7 (8.581) | -19.8 (8.474)
  Week 36: number analyzed (Participants) | 638 | 650
  Week 36 | -20.6 (8.439) | -19.7 (8.563)
  Week 40: number analyzed (Participants) | 632 | 649
  Week 40 | -20.5 (8.392) | -19.6 (8.393)
  Week 44: number analyzed (Participants) | 623 | 639
  Week 44 | -20.5 (8.384) | -19.6 (8.484)
  Week 48: number analyzed (Participants) | 625 | 638
  Week 48 | -20.5 (8.472) | -19.2 (8.509)
  Week 52: number analyzed (Participants) | 610 | 629
  Week 52 | -20.4 (8.301) | -19.2 (8.513)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Week 28; Test type: Superiority; p = 0.0489, ANCOVA; Least square mean (LSM) estimate = -0.09, 95% CI 2-sided [-0.18 to -0.00]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Week 32; Test type: Superiority; p = 0.1073, ANCOVA; LSM estimate = -0.09, 95% CI 2-sided [-0.19 to 0.02]
Statistical Analysis 3: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Week 36; Test type: Superiority; p = 0.0001, ANCOVA; LSM estimate = -0.24, 95% CI 2-sided [-0.37 to -0.12]
Statistical Analysis 4: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Week 40; Test type: Superiority; p = 0.0005, ANCOVA; LSM estimate = -0.25, 95% CI 2-sided [-0.38 to -0.11]
Statistical Analysis 5: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Week 44; Test type: Superiority; p = 0.0001, ANCOVA; LSM estimate = -0.30, 95% CI 2-sided [-0.45 to -0.15]
Statistical Analysis 6: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Week 48; Test type: Superiority; p = 0.0000, ANCOVA; LSM estimate = -0.49, 95% CI 2-sided [-0.70 to -0.27]
Statistical Analysis 7: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Test type: Superiority; p = 0.0000, ANCOVA; LSM mean = -0.59, 95% CI 2-sided [-0.81 to -0.36]

6. Secondary Outcome: Change From Baseline in PASI in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: as for outcome 5
Time Frame: Baseline, Weeks 28, 32, 36, 40, 44, 48 and 52
Population: Participants from the FAS-P75R, who had evaluable data at both baseline and the post-baseline time point, were analyzed. FAS-P75R: All participants who were rated as PASI 75 responders but did not achieve a PASI 90 response at Week 24, were randomized to treatment groups 3 or 4 and who received at least one dose of study drug at or after Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 114 | 92
score on a scale
  Week 28 | -16.1 (6.160) | -16.3 (8.029)
  Week 32: number analyzed (Participants) | 112 | 91
  Week 32 | -15.9 (6.002) | -16.6 (7.941)
  Week 36: number analyzed (Participants) | 111 | 92
  Week 36 | -16.1 (6.356) | -16.6 (7.996)
  Week 40: number analyzed (Participants) | 111 | 90
  Week 40 | -16.1 (6.908) | -16.8 (8.170)
  Week 44: number analyzed (Participants) | 108 | 89
  Week 44 | -16.1 (6.553) | -16.6 (8.259)
  Week 48: number analyzed (Participants) | 109 | 90
  Week 48 | -15.6 (6.246) | -16.8 (8.307)
  Week 52: number analyzed (Participants) | 104 | 90
  Week 52 | -15.5 (6.371) | -16.6 (8.011)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Week 28; Test type: Superiority; p = 0.1740, ANCOVA; LSM estimate = 0.40, 95% CI 2-sided [-0.18 to 0.99]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Week 32; Test type: Superiority; p = 0.0287, ANCOVA; LSM estimate = 0.79, 95% CI 2-sided [0.08 to 1.50]
Statistical Analysis 3: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Week 36; Test type: Superiority; p = 0.1202, ANCOVA; LSM estimate = 0.62, 95% CI 2-sided [-0.16 to 1.41]
Statistical Analysis 4: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Week 40; Test type: Superiority; p = 0.1157, ANCOVA; LSM estimate = 0.75, 95% CI 2-sided [-0.19 to 1.68]
Statistical Analysis 5: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Week 44; Test type: Superiority; p = 0.3189, ANCOVA; LSM estimate = 0.54, 95% CI 2-sided [-0.52 to 1.59]
Statistical Analysis 6: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Week 48; Test type: Superiority; p = 0.0240, ANCOVA; LSM estimate = 1.17, 95% CI 2-sided [0.16 to 2.18]
Statistical Analysis 7: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Week 52; Test type: Superiority; p = 0.0090, ANCOVA; LSM estimate = 1.47, 95% CI 2-sided [0.37 to 2.57]

7. Secondary Outcome: Change From Baseline in DLQI in Participants With a PASI 90 Response at Week 24
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral worts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment. A negative mean percentage change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: Only participants from the FAS-P90R, who had evaluable data at both baseline and week 52, were analyzed. The FAS-P90R included all participants who were rated as PASI 90 responders at the Week 24 visit, randomized to treatment groups 1 or 2 and received at least one dose of study drug at or after visit Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 605 | 624
score on a scale | -12.7 (7.325) | -11.4 (7.480)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Test type: Superiority; p = 0.0001, ANCOVA; LSM estimate = -0.62, 95% CI 2-sided [-0.93 to -0.31]

8. Secondary Outcome: Change From Baseline in DLQI in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 52
Population: Participants from the FAS-P75R, who had evaluable data at both baseline and week 52, were analyzed. FAS-P75R: All participants who were rated as PASI 75 responders but did not achieve a PASI 90 response at Week 24, were randomized to treatment groups 3 or 4 and who received at least one dose of study drug at or after Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 105 | 89
score on a scale | -10.0 (6.605) | -9.72 (6.880)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Test type: Superiority; p = 0.0675, ANCOVA; LSM estimate = 1.17, 95% CI 2-sided [-0.09 to 2.42]

9. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire - Psoriasis (WPAI-PSO) Score in Participants With a PASI 90 Response at Week 24
Description: The WPAI-PSO is a self-administered questionnaire comprised of 6 questions about effects of psoriasis on the patient's ability to work and perform regular activities based on the previous 7 days. The questionnaire quantifies the number of hours the respondent was unable to work and evaluates how much the respondent's psoriasis affected productivity while working. For respondents who were not in paid employment, the questionnaire evaluated how much the respondent's psoriasis affects their ability to perform regular daily activities. Four outcomes were generated from the WPAI-PSO: % Absenteeism: percent work time missed due to health; % Presenteism: percent impairment while working due to health; % Total work productivity impairment: percent overall work impairment due to health; % Total activity impairment: percent activity impairment due to health for all respondents. First 3 outcomes applied to employed participants only. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 644 | 662
score on a scale
  Absenteeism: number analyzed (Participants) | 360 | 356
  Absenteeism | -4.70 (19.590) | -1.99 (19.759)
  Presenteeism: number analyzed (Participants) | 361 | 348
  Presenteeism | -23.1 (25.968) | -23.0 (26.522)
  Total activity impairment: number analyzed (Participants) | 320 | 312
  Total activity impairment | -24.3 (27.850) | -23.2 (29.861)
  Work productivity loss: number analyzed (Participants) | 546 | 550
  Work productivity loss | -31.9 (29.392) | -28.6 (27.996)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Absenteeism; Test type: Superiority; p = 0.2101, ANCOVA; LSM estimate = -0.97, 95% CI 2-sided [-2.48 to 0.55]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Presenteeism; Test type: Superiority; p = 0.2971, ANCOVA; LSM estimate = -0.67, 95% CI 2-sided [-1.93 to 0.59]
Statistical Analysis 3: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Total activity impairment; Test type: Superiority; p = 0.5499, ANCOVA; LSM estimate = -0.61, 95% CI 2-sided [-2.59 to 1.38]
Statistical Analysis 4: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Test type: Superiority; p = 0.0758, ANCOVA; LSM estimate = -1.08, 95% CI 2-sided [-2.28 to 0.11]

10. Secondary Outcome: Change From Baseline in WPAI-PSO Score in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: as for outcome 9
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 114 | 92
score on a scale
  Absenteeism: number analyzed (Participants) | 54 | 49
  Absenteeism | -2.36 (12.990) | -3.45 (18.698)
  Presenteeism: number analyzed (Participants) | 52 | 48
  Presenteeism | -22.9 (28.377) | -22.1 (26.333)
  Total activity impairment: number analyzed (Participants) | 46 | 43
  Total activity impairment | -23.1 (28.657) | -21.7 (29.905)
  Work productivity loss: number analyzed (Participants) | 89 | 77
  Work productivity loss | -18.2 (28.824) | -22.5 (25.192)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Absenteeism; Test type: Superiority; p = 0.4156, ANCOVA; LSM estimate = 1.20, 95% CI 2-sided [-1.71 to 4.11]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Presenteeism; Test type: Superiority; p = 0.8619, ANCOVA; LSM estimate = 0.63, 95% CI 2-sided [-6.59 to 7.85]
Statistical Analysis 3: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Total activity impairment; Test type: Superiority; p = 0.6139, ANCOVA; LSM estimate = -0.61, 95% CI 2-sided [-6.31 to 10.61]
Statistical Analysis 4: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Work productivity loss; Test type: Superiority; p = 0.5674, ANCOVA; LSM estimate = 1.70, 95% CI 2-sided [-4.16 to 7.56]

11. Secondary Outcome: Change From Baseline in Pain, Itching and Scaling Score in Participants With a PASI 90 Response at Week 24
Description: Self-administered, 11-point numeric rating scales (NRS, 0-10) were used to evaluate the patients' assessment of their current pain, itching and scaling. Respondents answered the following questions for the assessment: Pain: Overall, how severe was your psoriasis-related pain over the past 24 hours?; Itching: Overall, how severe was your psoriasis-related itch over the past 24 hours?; and Scaling: Overall, how severe was your psoriasis-related scaling over the past 24 hours? Patients had to rate their pain, itching, and scaling from 0 to 10 (11-point scale), with the understanding that the 0 represents the absence or null end of the pain, itching, or scale intensity (i.e. no pain, itching or scaling) and the 10 represents the other extreme of pain, itching, or scaling intensity (i.e. pain, itching or scaling as bad as it could be). The number that the patient selected represents his or her intensity score in the respective category. A negative change from baseline indicates improvement
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 644 | 662
score on a scale
  Pain: number analyzed (Participants) | 495 | 478
  Pain | -4.56 (2.771) | -4.17 (2.2727)
  Itching: number analyzed (Participants) | 590 | 608
  Itching | -5.59 (2.885) | -5.20 (2.985)
  Scaling: number analyzed (Participants) | 598 | 610
  Scaling | -6.05 (2.659) | -5.73 (2.757)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Pain; Test type: Superiority; p = 0.1219, ANCOVA; LSM estimate = -0.13, 95% CI 2-sided [-0.30 to 0.04]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Itching; Test type: Superiority; p = 0.0001, ANCOVA; LSM estimate = -0.38, 95% CI 2-sided [-0.57 to -0.18]
Statistical Analysis 3: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Scaling; Test type: Superiority; p = 0.0003, ANCOVA; LSM estimate = -0.31, 95% CI 2-sided [-0.48 to -0.14]

12. Secondary Outcome: Change From Baseline in Pain, Itching and Scaling Score in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: as for outcome 11
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 114 | 92
score on a scale
  Pain: number analyzed (Participants) | 80 | 68
  Pain | -3.59 (2.754) | -3.68 (3.049)
  Itching: number analyzed (Participants) | 101 | 83
  Itching | -4.13 (2.883) | -4.49 (3.129)
  Scaling: number analyzed (Participants) | 102 | 89
  Scaling | -4.66 (2.960) | -5.40 (2.899)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Pain; Test type: Superiority; p = 0.6457, ANCOVA; LSM estimate = 0.17, 95% CI 2-sided [-0.57 to 0.92]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Itching; Test type: Superiority; p = 0.6136, ANCOVA; LSM estimate = 0.19, 95% CI 2-sided [-0.56 to 0.94]
Statistical Analysis 3: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Scaling; Test type: Superiority; p = 0.0203, ANCOVA; LSM estimate = 0.75, 95% CI 2-sided [0.12 to 1.39]

13. Secondary Outcome: Change From Baseline in the European Quality of Life - 5 Dimensions (EQ-5D) Visual Analogue Scale (VAS) in Participants With a PASI 90 Response at Week 24
Description: A visual analogue scale (VAS) was used within the EQ-5D. This scale recorded the respondent's self-rated health on a vertical 20-cm VAS where the endpoints were labeled "best imaginable health state" and "worst imaginable health state." This resulted in a numeric value set ranging from 0 (="worst imaginable health state") up to 100 (="best imaginable health state"). A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 603 | 620
score on a scale | 24.34 (23.296) | 21.24 (22.074)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Test type: Superiority; p = 0.0027, ANCOVA; LSM estimate = 2.22, 95% CI 2-sided [0.77 to 3.68]

14. Secondary Outcome: Change From Baseline in the EQ-5D VAS in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: A visual analogue scale (VAS) was used within the EQ-5D. This scale recorded the respondent's self-rated health on a vertical 20-cm VAS where the endpoints were labeled "best imaginable health state" and "worst imaginable health state." This resulted in a numeric value set ranging from 0 (="worst imaginable health state") up to 100 (="best imaginable health state").
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 103 | 88
score on a scale | 15.86 (20.099) | 18.92 (19.855)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Test type: Superiority; p = 0.2823, ANCOVA; LSM estimate = -2.31, 95% CI 2-sided [-6.55 to 1.92]

15. Secondary Outcome: Change From Baseline in the EQ-5D Utility Index (Germany, United Kingdom (UK)) in Participants With a PASI 90 Response at Week 24
Description: The EQ-5D quantifies the health state of a patient for the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort & anxiety/depression. In this study the EQ-5D-5L version has been used which evaluates each of these dimensions using the following 5 labels: no problems, slight problems, moderate problems, severe problems & unable to/extreme problems. Based on the 5 dimensions, a summary score (utility index) was derived using country specific value sets evaluating the patient condition described by the outcome in the single dimensions. The EQ-5D-5L (in this trail) utility index based on the crosswalk value sets available from the EuroQol for Germany & UK (https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/) was calculated. A positive change from baseline indicates improvement.
  A visual analogue scale was used within the EQ-5D measuring the health state of the patients, ranging from 0 (worst imaginable health state) up to 100 (best imaginable health state).
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 1 | Treatment Period 2: Group 2
Number analyzed (Participants) | 605 | 623
score on a scale
  Germany | 0.17 (0.200) | 0.13 (0.182)
  UK | 0.28 (0.250) | 0.22 (0.230)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; Germany; Test type: Superiority; p = 0.0861, ANCOVA; LSM estimate = 0.01, 95% CI 2-sided [-0.00 to 0.02]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 1 vs Treatment Period 2: Group 2; UK; Test type: Superiority; p = 0.0117, ANCOVA; LSM estimate = 0.02, 95% CI 2-sided [0.00 to 0.04]

16. Secondary Outcome: Change From Baseline in the EQ-5D Utility Index (Germany, UK) in Participants With a PASI Response of ≥75 to <90 at Week 24
Description: The EQ-5D quantifies the health state of a patient for the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. In the current study the EQ-5D-5L version has been used which evaluates each of these dimensions using the following five labels: "no problems", "slight problems", "moderate problems", "severe problems" and "unable to/extreme problems".
  Based on the five dimensions, a summary score (utility index) was derived using country specific value sets evaluating the patient condition described by the outcome in the single dimensions. For this trial, the EQ-5D-5L utility index based on the crosswalk value sets available from the EuroQol for Germany and for UK (https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/) was calculated.
  A visual analogue scale (VAS) was used within the EQ-5D measuring the health state of the patients, ranging from 0 (="worst imaginable health state") up to 100 (="best imaginable health state").
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
Number analyzed (Participants) | 103 | 89
score on a scale
  Germany | 0.11 (0.164) | 0.13 (0.164)
  UK | 0.18 (0.206) | 0.21 (0.204)
Statistical Analysis 1: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; Germany; Test type: Superiority; p = 0.1852, ANCOVA; LSM estimate = -0.02, 95% CI 2-sided [-0.05 to 0.01]
Statistical Analysis 2: Comparison: Treatment Period 2: Group 3 vs Treatment Period 2: Group 4; UK; Test type: Superiority; p = 0.2203, ANCOVA; LSM estimate = -0.03, 95% CI 2-sided [-0.07 to 0.02]

ADVERSE EVENTS:
Time Frame: Week 52
Description: The Adverse Events (AE) dataset has MedDRA version 19.1 (5345 records) and 20.0 (1272 records).
Arm/Group | Treatment Period 1: All Participants | Treatment Period 2: Group 1 | Treatment Period 2: Group 2 | Treatment Period 2: Group 3 | Treatment Period 2: Group 4
All-Cause Mortality (participants affected / at risk) | 1/1647 | 0/644 | 0/662 | 0/114 | 0/93
Serious Adverse Events (participants affected / at risk) | 73/1647 | 25/644 | 25/662 | 4/114 | 3/93
Other Adverse Events (participants affected / at risk) | 884/1647 | 272/644 | 288/662 | 64/114 | 60/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: All Participants (N=1647) | Treatment Period 2: Group 1 (N=644) | Treatment Period 2: Group 2 (N=662) | Treatment Period 2: Group 3 (N=114) | Treatment Period 2: Group 4 (N=93)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Giardiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 9 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 2 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 3 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Gastric cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Alcohol use (Social circumstances) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: All Participants (N=1647) | Treatment Period 2: Group 1 (N=644) | Treatment Period 2: Group 2 (N=662) | Treatment Period 2: Group 3 (N=114) | Treatment Period 2: Group 4 (N=93)
Vertigo (Ear and labyrinth disorders) | 4 | 2 | 2 | 1 | 2
Conjunctivitis allergic (Eye disorders) | 6 | 3 | 0 | 1 | 2
Eye pruritus (Eye disorders) | 5 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 74 | 16 | 22 | 4 | 0
Odynophagia (Gastrointestinal disorders) | 7 | 4 | 6 | 1 | 3
Toothache (Gastrointestinal disorders) | 34 | 11 | 11 | 3 | 1
Fatigue (General disorders) | 41 | 5 | 2 | 0 | 0
Injection site haematoma (General disorders) | 18 | 2 | 1 | 0 | 2
Pyrexia (General disorders) | 36 | 10 | 8 | 2 | 1
Bronchitis (Infections and infestations) | 23 | 12 | 6 | 1 | 3
Cystitis (Infections and infestations) | 12 | 3 | 3 | 0 | 2
Folliculitis (Infections and infestations) | 31 | 8 | 8 | 1 | 2
Gastroenteritis (Infections and infestations) | 22 | 10 | 10 | 3 | 2
Influenza (Infections and infestations) | 36 | 17 | 19 | 4 | 4
Nasopharyngitis (Infections and infestations) | 6 | 3 | 6 | 0 | 2
Oral candidiasis (Infections and infestations) | 25 | 9 | 14 | 0 | 3
Oral herpes (Infections and infestations) | 41 | 12 | 8 | 3 | 0
Pulpitis dental (Infections and infestations) | 4 | 1 | 2 | 2 | 2
Rhinitis (Infections and infestations) | 52 | 8 | 12 | 3 | 0
Sinusitis (Infections and infestations) | 22 | 8 | 6 | 1 | 2
Tonsillitis (Infections and infestations) | 34 | 8 | 9 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 65 | 18 | 16 | 7 | 5
Urinary tract infection (Infections and infestations) | 26 | 16 | 8 | 3 | 3
Viral upper respiratory tract infection (Infections and infestations) | 368 | 94 | 95 | 23 | 22
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 4 | 4 | 0 | 2
Alanine aminotransferase increased (Investigations) | 10 | 4 | 6 | 2 | 4
Aspartate aminotransferase increased (Investigations) | 8 | 4 | 3 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 | 16 | 19 | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 64 | 18 | 28 | 4 | 1
Headache (Nervous system disorders) | 141 | 31 | 27 | 6 | 1
Migraine (Nervous system disorders) | 9 | 1 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 61 | 11 | 10 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 46 | 13 | 17 | 3 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 9 | 4 | 1 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 20 | 8 | 14 | 3 | 1
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 65 | 9 | 11 | 2 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 21 | 12 | 16 | 11 | 8
Hypertension (Vascular disorders) | 55 | 7 | 10 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02409667/SAP_000.pdf
  • Study Protocol (2015-06-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT02409667/Prot_001.pdf